CLINICAL TRIAL: NCT02310607
Title: Non-invasive Optical Detection of Iron Deficiency - Evaluation of a Fiber Optic Tissue Fluorescence Measurement to Determine the Erythrocyte Zinc Protoporphyrin-IX/Heme Ratio
Brief Title: Non-invasive Optical Detection of Iron Deficiency
Status: Completed | Type: Observational
Sponsor: Klinikum der Universitaet Muenchen, Grosshadern (Other)
Responsible Party: Principal Investigator, Dr. Uwe Hasbargen, PD Dr. med., Klinikum der Universitaet Muenchen, Grosshadern
Other Study IDs: LFL_01/2012
Record Dates: First submitted 2014-12-02; First posted 2014-12-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Anemia, Iron-Deficiency
Keywords: Post-partum women
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Not an interventional study — Not an interventional study

SUMMARY:
This study aims to evaluate a prototype device detecting zinc protoporphyrin-IX fluorescence non-invasively from the intact oral mucosa. Zinc protoporphyrin-IX is an established indicator of iron deficiency. The prototype device is used to measure the erythrocyte zinc protoporphyrin-IX/heme ratio for women after delivery, a study group chosen because of an elevated risk of iron deficiency. The results from the non-invasive measurements are compared to reference measurements of the erythrocyte zinc protoporphyrin-IX/heme ratio from residual blood samples from the same patients and to other indicators of iron status, including hemoglobin, ferritin, serum iron, transferrin, transferrin saturation and soluble transferrin receptor.

Funding Source - Nestec Ltd.

DETAILED DESCRIPTION:
This trial is a proof-of-concept study using a prototype fiber optic fluorometer to acquire autofluorescence spectra from women after delivery and determine the erythrocyte zinc protoporphyrin-IX fluorescence intensity from these spectra. The non-invasively determined fluorescence spectra are evaluated to provide a quantitative measure of the erythrocyte zinc protoporphyrin-IX/heme concentration ratio. These values are primarily compared to an erythrocyte zinc protoporphyrin-IX determined by HPLC from residual blood samples from the same subjects and secondarily to erythrocyte zinc protoporphyrin-IX/heme ratios determined using a commercial hematofluorometer (AVIV, model 206d) and other indicators of iron status, including hemoglobin, ferritin, serum iron, transferrin, transferrin saturation and soluble transferrin receptor

This study could help to establish the non-invasive fluorescence measurement of zinc protoporphyrin-IX as a rapid, easy to use means for point-of-care screening for iron deficiency in resource-limited settings lacking laboratory infrastructure.

ELIGIBILITY:
Inclusion Criteria:

* Women after delivery of term infants
* Pregnancy and delivery without study-relevant complications
* Hb value pre-partum greater or equal 12 g/dL or less or equal 11 g/dL
* Regular blood withdrawal before and after delivery for clinical indications
* Informed consent to participation in the study
* Age 18 or older

Exclusion Criteria:

* Patients who are not legally competent
* Transfusion of blood products in the course of delivery
* Thalassemia and sickle cell anemia
* Any acute or chronic infectious or inflammatory disease
* Insufficient amount of residual blood in the clinically indicated post partum sample

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women post-partum
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2013-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Comparison of non-invasive erythrocyte zinc protoporphyrin IX measurements with HPLC reference (Spearman's Rho correlation, sensitivity and specificity) | 1 day after measurement
  Erythrocyte zinc protoporphyrin IX in the units of μmol/mol heme, as determined from non-invasive fluorescence and remission spectroscopic measurements at the oral mucosa, compared with reference standard determinations of erythrocyte zinc protoporphyrin IX in blood samples by high performance liquid chromatography (HPLC).

SECONDARY OUTCOMES:
Comparison of non-invasive erythrocyte zinc protoporphyrin IX measurements with estimate of body iron (sensitivity and specificity) | 1 day after measurement
  Erythrocyte zinc protoporphyrin IX in the units of μmol/mol heme, as determined from non-invasive fluorescence and remission spectroscopic measurements at the oral mucosa, compared with an estimate of total body iron, determined from the logarithm of the soluble transferrin receptor/ferritin ratio.

OTHER OUTCOMES:
Comparison of non-invasive erythrocyte zinc protoporphyrin IX measurements with hematofluorometer (Spearman's Rho correlation, sensitivity, specificity) | 1 day after measurement
  Comparison of non-invasive optical measurements of erythrocyte zinc protoporphyrin IX with determinations of erythrocyte zinc protoporphyrin IX in blood samples by commercial hematofluorometer.
Comparison of non-invasive erythrocyte zinc protoporphyrin IX measurements with hemoglobin (sensitivity and specificity) | 1 day after measurement
  Comparison of non-invasive optical measurements of erythrocyte zinc protoporphyrin IX with determinations of hemoglobin in blood samples.
Comparison of non-invasive erythrocyte zinc protoporphyrin IX measurements with ferritin (sensitivity and specificity) | 1 day after measurement
  Comparison of non-invasive optical measurements of erythrocyte zinc protoporphyrin IX with determinations of ferritin in blood samples.
Comparison of non-invasive erythrocyte zinc protoporphyrin IX measurements with serum iron (sensitivity and specificity) | 1 day after measurement
  Comparison of non-invasive optical measurements of erythrocyte zinc protoporphyrin IX with determinations of serum iron in blood samples.
Comparison of non-invasive erythrocyte zinc protoporphyrin IX measurements with transferrin (sensitivity and specificity) | 1 day after measurement
  Comparison of non-invasive optical measurements of erythrocyte zinc protoporphyrin IX with determinations of transferrin in blood samples.
Comparison of non-invasive erythrocyte zinc protoporphyrin IX measurements with transferrin saturation (sensitivity and specificity) | 1 day after measurement
  Comparison of non-invasive optical measurements of erythrocyte zinc protoporphyrin IX with determinations of transferrin saturation in blood samples.
Comparison of non-invasive erythrocyte zinc protoporphyrin IX measurements with soluble transferrin receptor (sensitivity and specificity) | 1 day after measurement
  Comparison of non-invasive optical measurements of erythrocyte zinc protoporphyrin IX with determinations of soluble transferrin receptor in blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Hasbargen, PD Dr. med., Principal Investigator — LMU Klinikum
Locations (1):
- Department of Obstetrics and Gynecology, Klinikum der Universitaet Muenchen, Grosshadern, Munich, Germany